CLINICAL TRIAL: NCT00995917
Title: A Randomized, Crossover, Pilot Trial of the Feasibility and Safety of Acupoint Injection of Vitamin K for Treatment of Primary Dysmenorrhea
Brief Title: A Pilot Study of Acupoint Injection for Primary Dysmenorrhea
Acronym: DAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A112809
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Dysmenorrhea; Pain, Menstrual
Keywords: acupuncture; menstrual pain; dysmenorrhea; menstrual cramps; vitamin K1
MeSH Terms: conditions — Dysmenorrhea | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin K acupoint injection (Experimental): Participants will receive the vitamin K intervention within 2 days of the onset of painful menstrual cramps.
  Interventions: Other: Vitamin K acupoint injection
- Saline Injection (Sham Comparator): Participants will receive the saline treatment within 2 days of the onset of painful menstrual cramps.
  Interventions: Other: Saline Injection

INTERVENTIONS:
Other: Vitamin K acupoint injection — Vitamin K will be injected into an acupuncture point within 2 days of the onset of painful menstrual cramps. Injections of 5 mg/0.5ml of vitamin K1 will be administered in bilateral acupuncture points. A single shot of vitamin K1 is 10mg/ml. Five mg/0.5ml will be drawn twice from one ampule and injected into each bilateral site, for a total dose of 10mg/ml of vitamin K.
  Arms: Vitamin K acupoint injection
Other: Saline Injection — Injection of .5ml saline bilaterally into both legs within 2 days of the onset of painful menstrual cramps.
  Arms: Saline Injection

SUMMARY:
Many women, particularly adolescent women, suffer from painful menstrual cramps, medically referred to as dysmenorrhea. Common treatments for menstrual cramps are non-steroidal anti-inflammatory drugs and oral contraceptives, but both have side effects that limit their use. Injection of vitamin K into an acupuncture point has been used as treatment for dysmenorrhea at the Obstetrics & Gynecology Hospital in Shanghai, China since at least 1985. More research is needed on the effectiveness of this treatment and its acceptability to different women. The objective of this study is to examine the feasibility and effectiveness of acupoint injection of vitamin K1 for the treatment of severe primary dysmenorrhea in the United States. Twenty participants will be randomized to receive either 1) vitamin K1 injection into an acupuncture point at the start of their menstrual cycle followed by a saline injection in a non-acupuncture point two months later or 2) saline injection in a non-acupuncture point followed by vitamin K1 injection into an acupuncture point two months later. The primary outcome measure will be change in pain intensity measured before and after each treatment. Data on other menstrual symptoms will be collected by telephone or a web-based survey. Three additional participants will be recruited to receive vitamin K1 injection into an acupuncture point and have blood samples drawn before and after injection to determine absorption of vitamin K1. The aims of the study are to collect preliminary data on the efficacy and safety of vitamin K1 injected in an acupoint for the treatment of severe primary dysmenorrhea; assess the feasibility and acceptability of the treatment among U.S. women; and test the blood absorption of vitamin K1 following acupoint injection treatment.

The investigators hypothesize that:

1. Vitamin K1 acupoint injection is a safe treatment for women with menstrual pain.
2. Vitamin K1 acupoint injection reduces menstrual pain more than placebo saline injection does.
3. The treatment of vitamin K1 acupoint injection is acceptable to U.S. women.
4. Vitamin K1 is absorbed into the blood thru acupoint injection.

ELIGIBILITY:
Inclusion Criteria:

* Young women age 18-25
* Severe primary dysmenorrhea (defined as severe, recurrent painful periods for 6 months or more, that are not due to any other diagnosis, and that have not been relieved, or have been only partially relieved by any other treatment)
* Nulliparous
* English speaking
* No acute or chronic conditions diagnosed or suspected
* Not on hormonal contraceptives
* Regular menstrual cycles for at least 6 months
* Has a working phone or pager

Exclusion Criteria:

* Use of hormonal contraceptives, or intra-uterine device
* Pregnancy
* Dysmenorrhea due to any other suspected or recognized causes
* History of abdominal surgery
* Participation in other concomitant therapy for acute or chronic pain
* Current treatment with anti-coagulant drugs for any reason
* Previous treatment with vitamin K acupoint injection
* Plans to be out of area during next 5 months
* Under age 18
* Known allergy to Vitamin K.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
self-reported pain | 3-5 months

SECONDARY OUTCOMES:
medications used during menstrual cycle | 3-5 months
activity restriction | 3-5 months
vitamin K content in blood | 1-2 months
Cox retrospective symptom scale | 3-5 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chao, Dr PH, MPA, Principal Investigator — University of California, San Francisco
Locations (1):
- Mount Zion Outpatient Unit, San Francisco, California, United States

REFERENCES:
- [Background] Davis AR, Westhoff CL. Primary dysmenorrhea in adolescent girls and treatment with oral contraceptives. J Pediatr Adolesc Gynecol. 2001 Feb;14(1):3-8. doi: 10.1016/s1083-3188(00)00076-0. PMID 11358700
- [Background] Milsom I, Minic M, Dawood MY, Akin MD, Spann J, Niland NF, Squire RA. Comparison of the efficacy and safety of nonprescription doses of naproxen and naproxen sodium with ibuprofen, acetaminophen, and placebo in the treatment of primary dysmenorrhea: a pooled analysis of five studies. Clin Ther. 2002 Sep;24(9):1384-400. doi: 10.1016/s0149-2918(02)80043-1. PMID 12380631
- [Background] Davis AR, Westhoff C, O'Connell K, Gallagher N. Oral contraceptives for dysmenorrhea in adolescent girls: a randomized trial. Obstet Gynecol. 2005 Jul;106(1):97-104. doi: 10.1097/01.AOG.0000165826.03915.65. PMID 15994623
- [Background] Yu J. Efficacy of vitamin K3 in the treatment of functional dysmenorrhoea: Clinical and laboratory observations. New Medicine and Clinical Trial. 1985:4
- [Background] Harlow SD, Park M. A longitudinal study of risk factors for the occurrence, duration and severity of menstrual cramps in a cohort of college women. Br J Obstet Gynaecol. 1996 Nov;103(11):1134-42. doi: 10.1111/j.1471-0528.1996.tb09597.x. PMID 8917003